CLINICAL TRIAL: NCT06115213
Title: Mass Screening of the Population of the North Kynouria Municipality in Arcadia, Greece for the Detection of Cardiovascular and Stroke Risk Factors
Brief Title: The North Kynouria Project
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Ioannina (Other)
Collaborators: Hellenic Stroke Organization (Unknown); Municipality of North Kynouria (Unknown); Greece 2021 Committee (Other Government); Astros Health Care Center (Unknown)
Responsible Party: Principal Investigator, Liontos Angelos, MD, MSc, PhD, University Hospital, Ioannina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: The North Kynouria Project
Record Dates: First submitted 2023-10-18; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Cerebrovascular Disease; Coronary Disease; Dyslipidemias; Stroke (CVA) or TIA; Myocardial Infarction; Hypertension; Diabetes Mellitus; Peripheral Artery Disease
Keywords: Atherosclerosis; Vascular Disease; Arterial Occlusive Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Cerebrovascular Disorders; Coronary Disease; Dyslipidemias; Stroke; Myocardial Infarction; Hypertension; Diabetes Mellitus; Peripheral Arterial Disease; Atherosclerosis; Vascular Diseases; Arterial Occlusive Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient screening (Experimental): Single group, no masking, receiving the intervention
  Interventions: Behavioral: Patient counselling

INTERVENTIONS:
Behavioral: Patient counselling — Patient counseling, lifestyle modifications, medication evaluation, and adherence
  Other Names: lifestyle modifications; dietary recommendations; smoking cessation; physical activity recommendations; medication adherence

SUMMARY:
The North Kynouria Project was initiated to study cardiovascular/stroke risk factors by employing mass screening and long-term surveillance of an adult population in the municipality of North Kynouria, in the county of Arcadia, Peloponnese, Greece. The North Kynouria Study was initiated to assess modifiable and non-modifiable determinants of cerebrovascular and coronary heart disease.

DETAILED DESCRIPTION:
BACKGROUND:

The North Kynouria Project is a longitudinal, interventional-behavioural, prospective study aiming to identify cardiovascular/stroke risk factors, in the adult population of the municipality of North Kynouria, in the county of Arcadia, Peloponnese, Greece. The project, initiated in November 2022, recruits volunteers, of both sexes, over 18 years of age, irrespective of their personal history of cardiovascular disease. The epidemiology and burden of cardiovascular disease in North Kynouria remain unknown. The study aims to explore and document the prevalence of major cardiovascular/stroke risk factors, as well as the nutritional status, cigarette smoking, exercise habits, alcohol consumption, and overall quality of life of the inhabitants.

DESIGN NARRATIVE:

The screening exam is conducted at the Astros, Health Center, by obtaining the patient's personal history, and information about the patient's habits, such as physical activity, smoking, and alcohol consumption. Body weight, height, and waist-to-hip ratio are also measured. During the examination, blood pressure is evaluated using a pre-specified protocol, including assessment of orthostatic hypertension. Further testing includes electrocardiography, ankle-brachial index, direct ophthalmoscopy, and carotid and cardiac ultrasound. Blood samples are collected and stored at the deep freeze of the Astros premises, and blood count, lipid panel, and liver and kidney function are measured.

The main field of interest is the prevalence and burden of risk factors and cardiovascular disease in the wider region of North Kynouria, Arcadia Greece. The project aims to assess the epidemiology of CVD and consequently improve public health and engage with the local community through healthy behavioral education.

ELIGIBILITY:
Inclusion Criteria:

* residents of North Kynouria

Exclusion Criteria:

* under 18,
* pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7000 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events | up to 5 years after enrollment
  myocardial infarction, ischemic and hemorrhagic stroke
All-cause mortality | up to 5 years after enrollment
  Death by any cause, cardiovascular, infection, cancer, other
Hospitalizations | up to 5 years after enrollment
  Any cause hospitalization
Emergency room visits | up to 5 years after enrollment
  Any cause of emergency room visit

SECONDARY OUTCOMES:
New diagnosis of Arterial hypertension | up to 1 year after enrollment
  Any diagnosis of arterial hypertension, masked, white-coat, nocturnal
New diagnosis of diabetes mellitus | up to 1 year after enrollment
  Type 1 or Type 2
New diagnosis of dyslipidemia | up to 1 year after enrollment
  New diagnosis or uncontrolled
New diagnosis of carotid atherosclerosis | up to 1 year after enrollment
  Evaluation of carotid artery stenosis
New diagnosis of peripheral artery disease | up to 1 year after enrollment
  Ankle Brachial Index evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Charalampos Milionis, MD, PhD, Principal Investigator — University of Ioannina; George Ntaios, MD, MSc, PhD, Principal Investigator — University of Thessaly
Locations (1):
- Astros Health Care Center, Ástros, Greece

IPD SHARING:
Plan to Share IPD: Yes
Study protocol details
Supporting Information: Study Protocol
Time Frame: 2024-2025
Access Criteria: Through access granting from the University of Ioannina